CLINICAL TRIAL: NCT03038659
Title: Predictive Value of Measuring Intima-media Thickness of Cavernosal Artery in Diagnosis of Arteriogenic Erectile Dysfunction by Penile Duplex
Brief Title: Role of Intima-media Thickness in Determining Arteriogenic Erectile Dysfunction
Status: Completed | Type: Observational
Sponsor: Adam International Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Raef Sadek, Dr. Ahmad Raef, Adam International Hospital
Other Study IDs: 2018
Record Dates: First submitted 2017-01-29; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Penile Duplex: Measuring intima media thickness
  Interventions: Device: Penile Duplex

INTERVENTIONS:
Device: Penile Duplex — Measuring intima media thickness

SUMMARY:
Erectile dysfunction.

DETAILED DESCRIPTION:
The intima media thickness is increasingly used as a surrogate end point of vascular outcomes in clinical trials aimed at determining the success of interventions that lower risk factors for atherosclerosis and associated diseases (stroke, myocardial infarction and peripheral artery diseases, like disease of cavernosal artery). The investigators hypothesized that the IMT of cavernosal artery would add to the predictive value of vasculogenic erectile dysfunction risk and outcomes. This study seeks to evaluate these hypotheses with our experience, investigating the predictive accuracy of Cavernosal Doppler ultrasound findings for discriminating patients with vasculogenic erectile dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* Erectile dysfunction patients

Exclusion Criteria:

* Penile trauma.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Erectile dysfunction pateints
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-29 (Actual)

PRIMARY OUTCOMES:
erectile dysfunction | six months
  intima media thickness

IPD SHARING:
Plan to Share IPD: No
Erectile dysfunction